CLINICAL TRIAL: NCT00424151
Title: Rituximab Treatment of Graves' Dysthyroid Ophthalmopathy Phase I/II
Brief Title: Rituximab Treatment of Graves' Dysthyroid Ophthalmopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Silkiss, Rona Z., M.D., FACS (Individual)
Collaborators: Lauer, Simeon, M.D. (Unknown); Reier, Alice M.D. (Unknown); Coleman, Morton M.D. (Unknown)
Responsible Party: Rona Z. Silkiss, MD, FACS, Rona Z. Silkiss, MD, FACS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U4126s
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Graves' Dysthyroid Ophthalmopathy; Thyroid Related Orbitopathy
Keywords: Graves' Disease; Dysthyroid Ophthalmopathy; Thyroid related orbitopathy
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This study is designed to treat patients with Graves' disease with Rituximab in an attempt to prevent or reverse the physically deforming and debilitating consequences of this disease.

DETAILED DESCRIPTION:
Graves' Dysthyroid ophthalmopathy is an autoimmune disease characterized by inflammatory changes of the periocular and orbital region often in association with an underlying thyroid abnormality. These changes can be extremely debilitating and may lead to visual loss. Attempts at limiting or reversing the phenotypic expression of Graves' ophthalmopathy through aggressive orbital decompression surgery or targeting the inflammatory disease, using high dose systemic corticosteroids and/or orbital radiotherapy, have been limited to date by treatment ineffectiveness and co-morbidities. Selective B-cell depletion therapy offers a potential treatment alternative. This study is designed to treat patients with Graves' disease with Rituximab in an attempt to prevent or reverse the physically deforming and debilitating consequences of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients eighteen years of age or older.Diagnosed with Graves' dysthyroid ophthalmopathy within one year of presentation.
* Manifest significant ophthalmic findings of active Graves' disease. (Clinical activity score 4 or greater)
* Evidence of thyroid abnormality (hyper or hypo thyroid) prior to thyroid treatment
* Elevated thyroid stimulating immunoglobulin, antithyroid peroxidase antibody or antithyroglobulin antibody.

Exclusion Criteria:

Long standing chronic disease. (greater than one year) History of ineffective prior orbital irradiation. Clinical activity score of less than 4.

* ANC < 1.5 x 103
* Hemoglobin: < 8.5 gm/dL
* Platelets: < 100,000/mm
* AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
* IgG: < 5.6 mg/dl and IgM: < .55 mg/dl
* Positive Hepatitis B or C serology (Hep B Surface antigen and Hep C antibody)
* History of positive HIV (HIV conducted during screening if applicable)
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera® / Rituxan®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical, mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation
* Concomitant malignancies or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac, including significant or uncontrolled arrhythmia, or pulmonary disease (including obstructive pulmonary disease)
* History of systemic lupus erythematosis
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.

Inability to comply with study and follow-up procedures

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Clinical response to treatment, alteration in immunoglobulin levels | One year post infusion
To assess the safety and tolerability of Rituximab in Graves' dysthyroid disease up to 24 weeks. Adverse and serious adverse events during the study period, reasonably or probably related to Rituximab, will be assessed at each study visit up to 12 month | One year
Efficacy: | One year after treatment
A significant (25%) reduction in progression of Thyroid Associated Ophthalmopathy or disease activity as measured by the thyroid associated ophthalmopathy scale (University of British Columbia Thyroid Orbitopathy Inflammatory Score) up to 24 weeks. | One year

SECONDARY OUTCOMES:
To evaluate for a reduction in disease activity as measured by: | One year
Reduction (25%) of elevated antibody levels- serum thyroid stimulating immunoglobulin (TSI), antithyroidperoxidase antibody (TPO) or antithyroglobulin levels at 24 weeks. | One year
MRI of the orbit with coronal and axial views to evaluate evidence of optic nerve crowding, muscle size reduction or decreased proptosis during treatment and follow up interval at 24 weeks. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Rona Z Silkiss, MD, Principal Investigator — California Pacific Medical Center
Locations (2):
- United States (2):
  - Rona Z. Silkiss, MD, FACS, Oakland, California
  - Simeon A. Lauer, MD, New York, New York